CLINICAL TRIAL: NCT01106963
Title: Nail Position Has an Influence on Anterior Knee Pain After Tibial Intramedullary Nailing
Brief Title: Anterior Knee Pain After Tibial Nailing
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: General Hospital Varazdin, National Health Insurance
Other Study IDs: AKP
Record Dates: First submitted 2010-04-14; First posted 2010-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Knee Pain
Keywords: knee; tibial fractures; pain; osteosynthesis; intramedullary nailing
MeSH Terms: conditions — Tibial Fractures; Pain | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tibial shaft fractures: Patients had tibial shaft fractures in the last 3 years. All were treated with intramedullary (IM) reamed nails with 2 or 3 interlocking screws.
  Interventions: Procedure: Tibial intramedullary nailing

INTERVENTIONS:
Procedure: Tibial intramedullary nailing — Patients' operations were performed using the peritendinous approach. A medial longitudinal incision was made, with care being taken not to damage the patellar tendon or its sheath. Standard proximal and distal locking screws were used. All patients were given postoperative instructions for thigh muscle rehabilitation and the same physiotherapy was performed after IM nailing during hospitalization. Nails were removed from some of the patients with the presence of knee pain or pain at the insertion points of the locking screws, however, no nails were removed earlier than one year postoperatively. Proof of the healed bone fracture was confirmed by radiologic examination.
  Other Names: tibial fractures; intramedullary nailing

SUMMARY:
Anterior knee pain (AKP) is a common complication following intramedullary (IM) nailing of a tibial shaft fracture. The purpose of this prospective study was to determine if there is an association between AKP and nail position. The investigators have analyzed postoperative outcome results and the possible relationship between AKP according to the visual-analog scale (VAS) scale, and nail position marked as a distance from the tip of the nail to the tibial plateau (NP) and tuberositas tibiae (NT), measured postoperatively on L-L knee X-rays.

DETAILED DESCRIPTION:
The aim of this study was to determine the possible relationship between anterior knee pain (AKP) and nail position marked as a distance from tip of nail to tibial plateau (NP) and to the tuberositas tibiae (NT).

We evaluated postoperative outcome results of 50 patients in the last 3 years with healed fractures initially treated with intramedullary (IM) reamed nails with 2 or 3 interlocking screws on both parts of the nail and with the use of medial peritendinous incision for nail entry portal. Patients marked a point on the visual analog scale (VAS) that corresponded to the level of postoperative AKP felt. Two groups of patients were formed on the basis of AKP (pain level was neglected): groups A and B, with and without pain, respectively.

We found that the difference between the two groups concerning NP measurements was statistically significant, but not concerning NT measurements (P < 0.05). Patients were classified by pain with high accuracy (98%) according to a classification tree.

We conclude that the symptoms of AKP did not appear if the tip of the nail position was more than 6.0 mm from the NP and more than 2.6 mm from the NT. However, for better evaluation of these results it will be necessary to examine more postoperative patients with AKP.

ELIGIBILITY:
Inclusion Criteria:

* tibial shaft fractures
* fracture treatment with intramedullary nailing with 2 or 3 interlocking screws on both ends of the nail

Exclusion Criteria:

* amputated legs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of primary care hospital trauma patients with tibial shaft fractures treated with intramedullary nailing.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Anterior knee pain | 1 year
  Anterior knee pain was assessed postoperatively with the visual analog scale (VAS). Patients generally had pain when kneeling, at the insertion point of surgical screws, or at the back of knee upon flexing.

CONTACTS AND LOCATIONS:
Overall Officials: Nikica Darabos, MD, PhD, Principal Investigator — University of Zagreb School of Medicine
Locations (1):
- University of Zagreb School of Medicine, Department of Traumatology, Zagreb, Croatia